CLINICAL TRIAL: NCT04264325
Title: Quantitative Diaphragmatic Ultrasound Evaluation in Pleural Effusions
Brief Title: Quantitative Diaphragmatic Ultrasound Evaluation in Pleural Effusions : A Feasability Study
Acronym: ADD-Echo
Status: Completed | Type: Observational
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Other Study IDs: 7565
Record Dates: First submitted 2020-01-30; First posted 2020-02-11 (Actual); Last update posted 2023-05-10 (Actual); Status verified 2023-05

CONDITIONS: Malignant Pleural Effusion; Lung Neoplasms
Keywords: Dyspnea; Malignant pleural effusion; Lung Neoplasms; Therapeutic thoracocentesis; Lung ultrasound; Diaphragmatic ultrasound; Diaphragmatic dysfunction
MeSH Terms: conditions — Pleural Effusion, Malignant; Lung Neoplasms; Dyspnea

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Malignant pleural effusions : diaphragmatic ultrasound measure
  Interventions: Other: diaphragmatic ultrasound measure

INTERVENTIONS:
Other: diaphragmatic ultrasound measure — patients with lung neoplasms and malignant pleural effusions who need a diagnostic or therapeutic thoracocentesis

SUMMARY:
Malignant pleural effusions cause breathlessness and impairs quality of life. Thoracocentesis is frequently used to relieve breathlessness.

The severity of breathlessness correlates poorly with the size of the effusion. Symptom reduction from fluid drainage varies between patients. No predictors exist to identify which patients benefits more of pleural effusion. One study suggests that a inverted hemidiaphramatic (inverted shape) is associated with a greater dyspnea improvement. Others parameters of diaphragmatic motion have not been studied till now.

This study aims to evaluate the feasability of diaphragmatic ultrasound evaluation (shape by B-mode, quiet, deep inspiratory motion and sniff diaphragm motion by TM-mode) before and after pleural drainage.

Primary end point aims to evaluate the feasability of deep breath inspiratory excursion in ipsilateral side of thoracocentesis by anterior subcostal approach in the mid-clavicular line in the right in patients with malignant pleural effusions. The liver or spleen was identified as a window for each hemidiaphragm.

Secondary end points aim to evaluate

* the feasability of quiet breath inspiratory motion ,
* the feasability of sniff diaphragm motion
* the feasability of deep breath inspiratory motion by posterior method
* the comparaison of feasibility with different types of breathing and or anterior or posterior approach for ultrasound
* the feasability of the shape by B-mode.
* the correlation between the change of the shape of ipsilateral diaphragm and the evolution of dyspnea, before and after thoracocentesis.
* the correlation between the volume of pleural effusion evacuated and the evolution of dyspnea, before and after thoracocentesis.
* the comparaison of the changing of dyspnea in patients with noticed paradoxal movement of diaphragm before thoracocentesis and patients with persistent paradoxal/or non persistant paradoxal movement of ipsilateral hémidiaphragm.
* the correlation between the feasability of diaphragmatic ultrasound motion measurments evaluation and the body mass index.
* the comparaison between the different diaphragmatic ultrsound times for anterior or posterior approach.

ELIGIBILITY:
Inclusion Criteria:

* Age> 18 years old
* Male or female patient
* Patient with known lung cancer, regardless of histology or suspected of having unknown lung cancer or relapse / progression of lung cancer
* Presenting a pleural effusion with clinical necessity of evacuating pleural puncture
* Subject who expressed his non opposition to the research

Exclusion Criteria:

* Patient's refusal to participate in the study
* History of pleurodesis whatever the indication (pneumothorax or recurrent pleural effusion) or the technique used
* Permanent chest drain
* inability to provide informed information to the subject (subject in an emergency, difficulty understanding the subject, etc.)
* Subject under judicial protection
* Subject under guardianship or curatorship
* Pregnant or lactating woman

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 30 patients with lung neoplasms and malignant pleural effusions who need a diagnostic or therapeutic thoracocentesis
Sampling Method: Non-Probability Sample
Enrollment: 15 (Actual)
Dates: Start 2020-01-31 (Actual); Primary Completion 2020-08-20 (Actual); Study Completion 2023-05-03 (Actual)

PRIMARY OUTCOMES:
Evaluate the feasibility of measuring the diaphragmatic amplitude in wide breathing (RA) on the side homolateral to the pleural puncture | one day
  Rate of patients with a feasible measure of diaphragmatic amplitude in wide breathing (RA), on the side homolateral to the pleural puncture, by the anterior route before and after pleural puncture.

SECONDARY OUTCOMES:
Feasability of quiet breath inspiratory motion | one day
  Rate of patients with a feasible measure of diaphragmatic amplitude in spontaneous breathing (RS), on the side homolateral to the pleural puncture, by the anterior route before and after pleural puncture.

CONTACTS AND LOCATIONS:
Overall Officials: Mickaël OHANA, Principal Investigator — Hôpitaux Universitaires de Strasbourg
Locations (1):
- Les Hôpitaux Universitaires de Strasbourg, Strasbourg, France

IPD SHARING:
Plan to Share IPD: Undecided